CLINICAL TRIAL: NCT07165444
Title: Potassium-Competitive Acid Blocker Versus Proton Pump Inhibitor as A Part of Bismuth Based Quadruple Therapy for Treatment of Helicobacter Pylori Infection: A Randomized Controlled Trial
Brief Title: Potassium-Competitive Acid Blocker Versus Proton Pump Inhibitor as A Part of Bismuth Based Quadruple Therapy for Treatment of Helicobacter Pylori Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Galal Flefel, Lecturer of Internal Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR1285/7/25
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Potassium-Competitive Acid Blocker; Proton Pump Inhibitor; Bismuth Based Quadruple Therapy; Treatment; Helicobacter Pylori Infection
MeSH Terms: interventions — Proton Pump Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B-CAP group (Experimental): Patients will a 10-day course of bismuth, metronidazole, tetracycline four times daily, and vonoprazan 20 mg twice daily.
  Interventions: Drug: Potassium-Competitive Acid Blocker
- PPI group (Active Comparator): Patients will receive a 10-day course of bismuth, metronidazole, tetracycline four times daily, and rabeprazole 20 mg twice daily.
  Interventions: Drug: Proton Pump Inhibitor

INTERVENTIONS:
Drug: Potassium-Competitive Acid Blocker — Patients will a 10-day course of bismuth, metronidazole, tetracycline four times daily, and vonoprazan 20 mg twice daily.
  Arms: B-CAP group
Drug: Proton Pump Inhibitor — Patients will receive a 10-day course of bismuth, metronidazole, tetracycline four times daily, and rabeprazole 20 mg twice daily.
  Arms: PPI group

SUMMARY:
This study aims to compare the eradication rate, safety, and patient adherence between potassium-competitive acid blockers (P-CABs) and proton pump inhibitor-based bismuth quadruple therapy in patients with Helicobacter pylori infection.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a spiral-shaped, Gram-negative bacterium that colonizes the stomach lining and is considered one of the most prevalent chronic infections globally.

Bismuth-based quadruple therapy (proton pump inhibitor, bismuth, metronidazole, and tetracycline) is considered an effective alternative in cases of antibiotic resistance. This regimen achieves high eradication rates, even in areas with dual clarithromycin and metronidazole resistance.

Potassium-competitive acid blockers (P-CABs), such as vonoprazan, provide rapid, consistent, and strong acid suppression regardless of the CYP2C19 genotype.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Both sexes.
* Confirmed Helicobacter pylori infection by stool antigen (3rd-gen ELISA) or urea breath test (UBT).
* No prior eradication therapy.

Exclusion Criteria:

* Prior Helicobacter pylori treatment.
* Use of antibiotics, proton pump inhibitor, or bismuth in the prior 4 weeks.
* Gastric surgery history.
* Major organ failure.
* Pregnancy or lactation.
* Known allergy to study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | 2 weeks after proton pump inhibitor
  Helicobacter pylori eradication rate will be recorded.

SECONDARY OUTCOMES:
Adverse drug reactions | 2 weeks after proton pump inhibitor
  Adverse drug reactions will be recorded.
Patient adherence | 2 weeks after proton pump inhibitor
  Adherence will be assessed by asking patients to return used packaging and by questioning.
Degree of patient satisfaction | 2 weeks after proton pump inhibitor
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.